CLINICAL TRIAL: NCT00164489
Title: Intervention Research Grants to Promote the Health of People With Disabilities
Brief Title: Health Promotion of People With Disabilities
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCBDDD-CCR523273
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid and Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Behavioral: Weight control and physical activity promotion

SUMMARY:
This research is meant to evaluate the effectiveness of two different prevention programs for post-acute management of rheumatoid and osteo-arthritis

DETAILED DESCRIPTION:
Park Nicollet Clinic and the Institute for Clinical Systems Integration (ICSI) have developed evidence-based care guidelines and intervention strategies including degenerative joint disease. Included in these guidelines are risk factors for increased limitations, obesity and physical activity.

The aims of this research are to modify well-established weight management techniques and physical activity promotion interventions according to ICSI recommendations, implement the interventions in a diverse patient population, demonstrate the short and long term impact of the interventions.

The approach will be an individual randomized controlled trial of 400 patients, 200 each in a coach-supported intervention, 200 in a self-directed intervention.

ELIGIBILITY:
Inclusion Criteria:

* clinical visit 11/1/2003 to april 30/2004 diagnosis code rheumatoid arthritis or lower extremity osteoarthritis saw a provider that consented to have patients invited to participate consented to being contacted for research

Exclusion Criteria:

-

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2003-10; Study Completion 2005-06

PRIMARY OUTCOMES:
height weight: BMI
Healthy physical activity levels: 20 minutes of physical activity 4+ days/week

SECONDARY OUTCOMES:
improved weight status
improved diet
decreased pain
reduced depression

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Braun, Ph.D., Principal Investigator — HealthPartners Institute
Locations (1):
- Park Nicollet Institute, Minneapolis, Minnesota, United States